CLINICAL TRIAL: NCT04483388
Title: Training With Virtual Reality in Upper Arm Reaching of Children With Cerebral Palsy: Crossover Randomized Clinical Trial
Brief Title: Training With Virtual Reality in Upper Arm Reaching of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Natália Feitoza do Nascimento, Clinical Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12649913.0.0000.5537
Record Dates: First submitted 2015-08-11; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2015-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Rehabilitation; Physiotherapy; Virtual Reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group AB (Other): After randomization, 6 children composed the AB sequence were initially submitted to experimental training with virtual reality and after a week, a period considered washout, the conventional training.
  Interventions: Other: Training with Virtual Reality; Other: Conventional Training
- Group BA (Other): After randomization 6 children composed the BA sequence were initially submitted to conventional training and after a week, a period considered washout, the experimental training with virtual reality.
  Interventions: Other: Training with Virtual Reality; Other: Conventional Training

INTERVENTIONS:
Other: Training with Virtual Reality — Computed virtual reality therapy was performed using the Nintendo Wii® console equipment. This system allows interaction with the player by means of a movement detection system and the representation of his avatar graphical representation of a user in virtual reality. It has a remote control with a wireless system, responsible for capturing the speed, direction , acceleration and deceleration of movement. The movements performed by the player are captured and reproduced on a screen via an infrared light sensor, positioned above the TV. The feedback given by the TV provides the movement itself observing opportunity in real time, generating positive reinforcement and facilitating training and improved task. The software used in this study was the Nintendo Wii Sports.
  Other Names: Training A
Other: Conventional Training — It was done five types of exercises following to the protocol:
  Exercise 1 (shoulder abduction); Exercise 2 (external rotation of the shoulder); Exercise 3 (elbow extension); Exercise 4 (weight transfer in upper limbs: a sitting position); Exercise 5 (function: task-oriented training).
  Other Names: Training B

SUMMARY:
The objective of this study was to evaluate the effects of training with Virtual Reality in the movement range of children with Cerebral Palsy spastic hemiparetic.The study protocol consisted of two days of training and 1 revaluation. The training A (Nintendo Wii®) and B (standard protocol) were randomized the children in AB and BA sequences, with one week interval. Immediately kinematics pre and post-training was held and after a week no significant changes were observed for the angular variables and space-time between groups. The Virtual Reality used for intervention to improve upper arm function in children with Cerebral Palsy is still a relatively new method.

DETAILED DESCRIPTION:
Introduction: The disability of upper limb function (MS) of children with Cerebral Palsy (CP) spastic hemiparetic restricts their participation in social activities. Virtual reality (VR) has shown promising results in functional recovery of this population, however, few studies have evaluated its effectiveness in the reaching of motion of these children. Objective: To assess the effects of training with VR in the movement range of children with CP spastic hemiparetic. Materials and Methods: We conducted a randomized crossover trial, where the sample consisted of 12 children diagnosed with CP hemiparetic, both genders, with a mean age of 9.63 ± 2.3 years. The sample description was performed by assessing muscle tone, range of motion, grip strength, functional performance and disability. Kinematic analysis of the upper limb was performed by Qualisys Motion Capture System®. The study protocol consisted of two days of training and 1 revaluation. The training A (Nintendo Wii®) and B (standard protocol) were randomized the children in AB and BA sequences, with one week interval. Immediately kinematics pre and post-training was held and after a week. Data were analyzed using SPSS 20.0 (Statistical Package for Social Science) assigning a 5% significance level. The kinematic variables were analyzed by two-way ANOVA for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cerebral palsy spastic hemiparesis;
* Aged 6 to 12 years old;
* Preserved cognition to understand instructions;
* Present no significant auditory and visual deficits;
* The affected upper limb classified in levels II and III Rating System Manual (MACS, English Manual Abilities Classification System). The level II corresponds to children who are able to handle the majority of objects with low quality and / or speed of movement, while at level III are those that manipulate objects with difficulty and low speed, requiring assistance organization of activity. Spasticity ranked among the levels 0 and 3 of the Modified Scale Ashworth.It has not performed orthopedic surgeries, or have made use of botulinum toxin for less than six months, not presenting seizures, controlled medication.

Exclusion Criteria:

* Presence of pain or discomfort during the course of the training;
* Refusal to follow commands and instructions and discontinuity of interventions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Kinematic upper arm evaluation of children with cerebral palsy | 4 months
  We used a standardized 3D-analysis protocol to evaluate upper limb kinematic. The evaluation was divided into two stages: static collection and dynamics. In static collection, the patient was seated on a bench with feet on the floor, so that a 90 ° angle hip, knee and ankle joints. A table was positioned at a distance of 100% of the length of the affected upper arm and at the height of the xiphoid process and were used 19 mm reflective markers at the following points anatomical. In the dynamic evaluation, the participant continued to sit on the bench, with arms at the side of the torso, maintaining 90 ° elbow flexion and hand on the table was asked to touch a cube. All children started reach movement with the unaffected limb. Therefore, 15 reaches per child in each member in total and it was performed one minute intervals between attempts. The following variables: duration of movement, peak velocity and angular variation of shoulder and elbow.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Raquel Lindquist, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte

REFERENCES:
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Siebes RC, Wijnroks L, Vermeer A. Qualitative analysis of therapeutic motor intervention programmes for children with cerebral palsy: an update. Dev Med Child Neurol. 2002 Sep;44(9):593-603. doi: 10.1017/s0012162201002638. PMID 12227614
- [Background] Coleman A, Weir KA, Ware RS, Boyd RN. Relationship between communication skills and gross motor function in preschool-aged children with cerebral palsy. Arch Phys Med Rehabil. 2013 Nov;94(11):2210-7. doi: 10.1016/j.apmr.2013.03.025. Epub 2013 Apr 11. PMID 23583864
- [Result] Wu WC, Hung JW, Tseng CY, Huang YC. Group constraint-induced movement therapy for children with hemiplegic cerebral palsy: a pilot study. Am J Occup Ther. 2013 Mar-Apr;67(2):201-8. doi: 10.5014/ajot.2013.004374. PMID 23433275
- [Result] Chen YP, Kang LJ, Chuang TY, Doong JL, Lee SJ, Tsai MW, Jeng SF, Sung WH. Use of virtual reality to improve upper-extremity control in children with cerebral palsy: a single-subject design. Phys Ther. 2007 Nov;87(11):1441-57. doi: 10.2522/ptj.20060062. Epub 2007 Sep 25. PMID 17895352
- [Result] Chiu HC, Ada L, Lee HM. Upper limb training using Wii Sports Resort for children with hemiplegic cerebral palsy: a randomized, single-blind trial. Clin Rehabil. 2014 Oct;28(10):1015-24. doi: 10.1177/0269215514533709. Epub 2014 May 21. PMID 24849793
- [Result] Chen YP, Lee SY, Howard AM. Effect of virtual reality on upper extremity function in children with cerebral palsy: a meta-analysis. Pediatr Phys Ther. 2014 Fall;26(3):289-300. doi: 10.1097/PEP.0000000000000046. PMID 24819682